CLINICAL TRIAL: NCT01708031
Title: Computerized Mental Arthimetic Task Based Human Stress Level Detection Using Physiological Signal
Acronym: UNIMAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universiti Malaysia Perlis (Other)
Responsible Party: Principal Investigator, KARTHIKEYAN PALANISAMY, Mr, Universiti Malaysia Perlis
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: MAT STRESS
Record Dates: First submitted 2012-10-10; First posted 2012-10-16 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Stress, Psychological
MeSH Terms: conditions — Stress, Psychological | interventions — Skin Temperature

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- stress inducing task (Experimental): Normal subjects without history medication presently will be participated. Stress induced through stress inducing task (mental arithmetic task), the physiological signals collected before and during the task simultaneously. All the subjects will be participating only once in this MAT based study. Because, the stress will not be possible to induce when the subject is more familiar with the stress inducing task.
  Interventions: Other: physiological signals

INTERVENTIONS:
Other: physiological signals
  Other Names: ECG; EMG; GSR; Skin temperature; EEG; BP

SUMMARY:
Computerized Mental Arithmetic Task Based Human Stress Level Detection Using Physiological Signal

The objective of this study is to induce and measure the human stress level through computerized mental arithmetic task and multiple physiological signals (ECG, EMG, GSR, and skin temperature). Studies suggested that mental arithmetic task is one of the efficient stimuli to induce the stress. Hence, this mental arithmetic task protocol has been improved in to computerized version. The protocol will be tested with normal subjects and multiple physiological signals will be acquired simultaneously. The questionnaire about the subject experience will be obtained in order to strengthen the stress induction. The normal volunteer subjects will be invited for the participation this study. The physiological signal will be analyzed using suitable algorithm based on the characteristics of each signals. The multiple signal based stress level assessment system will be developed by training and testing the acquired data.

DETAILED DESCRIPTION:
Mental arithmetic task (MAT) is frequently used stressor to induce and assess stress by efficiently. However, this method not standardized until today, it is due to different environmental and psychological factors on the experimental condition. Different protocol designs used in various stress assessment studies are elaborated

Previous protocol details using MAT based stress induction

(Lundberg & Melin, 1994) 62 subjects & SBP (Systolic Blood Pressure), DBP (Diastolic Blood Pressure), Heart rate and EMG.

* A series of addition and subtraction of 1 digit numbers.
* Subject pronounces the answer and errors will be recorder by tape recorder.
* Soft music was played to relax the subject and physiological and psychological parameters were measured.

(Ushiyama, et al., 1991) 26 subjects, blood samples, BP and ECG. Initially, 20 minute relaxation

* 7 subtractions from 700 within 2.5 min after the relaxation. Finally 3 minute relaxation.
* ECG continuous measure for complete duration
* Blood samples, blood pressure for discrete variable only once on each task.

(Tomaka, Blascovich, & Swart, 1994b) 41 subjects & heart rate, skin conductance response (SCR), stroke volume (SV), SBP and DBP

* Mental arithmetic task with two type, with silent phase, and aloud phase.
* Initially, 10 minute rest before electrode placement and 4 minutes relaxation after the electrode placement and calibration.
* Type1, rapid serial addition by 13 from 2549. Duration 4 minutes with 5 minute final relaxation.
* Type 2, rapid serial subtraction by 7 from 2549. Duration 4 minutes with 5 minute final relaxation.
* The subject is vocalizing the answer in a loud phase and silent phase subject to be silent and should perform the task.

(Ring, Drayson, Walkey, Dale, & Carroll, 2002) 24 subjects & SBP, DBP and pulse rate.

* 4 seven minute series addition with presentation rate of 3.5, 3.0, 2.5 and 2.0s respectively.
* Addition of two sequentially presented single digit numbers (from1 to 9) in audio.
* Answers should be retained in the memory for next addition that presented on the audio tape recorder.
* SBP, DBP and pulse rate is a discrete variable taken from a certain interval of time.

(Linden, 1991) 61 subjects & DBP, SBP heart rate.

* Four different kind noise distraction during MAT. Subtraction of 2000 from 6,7, 8,9 consecutively, calculation time is 5 Sec per one step.
* Verbally pronounce the answer.
* No noise task (the task performed without any noise).
* Variable real life noise ( siren, car engine warm up, thunder getting closer, background noise of train station etc.,).
* Steady real life noise (coffee and bar shop background noise).
* Variable meaningless noise task(white and pink noise).

(Von Dawans, Kirschbaum, & Heinrichs, 2010) 25 subjects & ECG

* Mental arithmetic task (serial subtraction) of 8 min.
* The task performed in between other stress inducing task.

(Seraganian, Szabo, Brown, & Behavior, 1997) 20 subjects & ECG.

* 11 problems requiring two serial arithmetic operations with integers (e.g., 14* 6-17).
* Subject should perform arithmetic and also rate the difficulty level 10 point scale.
* Task were presented in tape recorder in counter balanced order
* Heart rate was continues measure.

Protocol design information

In this work, MAT is designed to induce and increase the stress level from one level to another by creating and increasing mental demand from easy to hard. Here, the mental arithmetic task is designed with audio distraction to reduce the cognition while in mental demand or load. This continuous exposure is reason to induce the stress of the participants. The protocol consist of 4 different levels such as relaxation with soft music, low level (low difficulty), medium level (medium difficulty), high level (high difficulty). Each level has 30 arithmetic problem addition, subtraction, multiplication and division or combination of these. Complexities of problem between levels are designed according to the low, medium, and high. 10 randomly selected real time noises (generator, siren, motor sound etc) are added with every 10 problems of each level in order to reduce the concentration and increase the mental demand. According to the data collection environment, the noises are calibrated and controlled.

Physiological measures

Non-intrusive measurement Electrocardiogram Electromyogram Galvanic skin response Skin temperature Electroencephalogram

Subject information

Normal subjects and open invitation will be given to select the volunteers

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

- no histroy of disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-04 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Stress levels assesment desinged based on the physiological signal acquired from the various subject by using MAT protocal. | 90 minutes
  Selection of physiological signals
  The following four physiological signal will be acquired based on the strong clinical evidence, Non-intrusive measurement, and futuristic to develop the real time detection system using compact electronics that to reduce the obtrusive of the human in real time activities such as in job, sports application.
  Electromyogram Galvanic skin response Skin temperature

CONTACTS AND LOCATIONS:
Overall Officials: Sazali Yaacob, PhD, Principal Investigator — Unimap; Murugappan M, PhD, Study Chair — Unimap
Locations (1):
- Unimap, Kangar, Perlis, Malaysia